CLINICAL TRIAL: NCT02898142
Title: Evaluation of Intestinal and Hepatic Parts in Fasting Postprandial Hypertriglyceridemia in Patients With or Without Metabolic Syndrome
Brief Title: Intestines and Liver Contribution to Fasting Postprandial Hypertriglyceridemia
Acronym: TRIGPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P111003
Record Dates: First submitted 2015-12-21; First posted 2016-09-13 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2015-12

CONDITIONS: Hypertriglyceridemia; Metabolic Syndrome
Keywords: Postprandial test; Metabolic syndrime; HTG
MeSH Terms: conditions — Hypertriglyceridemia; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isolated HTG without metabolic syndrome (Experimental): Postprandial test : The preparation used for this test consists of a semi standardized liquid meal (400 ml energy drink Fresubin® 2 cal / ml, Fresenius Kabi, France), containing 800 kcal, 50% calories from carbohydrates, 15% in as protein, and 35% as lipid. The test meal will be performed in the morning during 6 hours (between 8:00 and 14:00) after 10 hours of fasting.
  Interventions: Other: Postprandial test
- HTG with metabolic syndrome (Experimental): Postprandial test : The preparation used for this test consists of a semi standardized liquid meal (400 ml energy drink Fresubin® 2 cal / ml, Fresenius Kabi, France), containing 800 kcal, 50% calories from carbohydrates, 15% in as protein, and 35% as lipid. The test meal will be performed in the morning during 6 hours (between 8:00 and 14:00) after 10 hours of fasting.
  Interventions: Other: Postprandial test

INTERVENTIONS:
Other: Postprandial test — Postprandial test : The preparation used for this test consists of a semi standardized liquid meal (400 ml energy drink Fresubin® 2 cal / ml, Fresenius Kabi, France), containing 800 kcal, 50% calories from carbohydrates, 15% in as protein, and 35% as lipid. The test meal will be performed in the morning during 6 hours (between 8:00 and 14:00) after 10 hours of fasting. This post prandial test is the same in the two study groups.

SUMMARY:
Fasting and postprandial hypertriglyceridemia (HTG) depends on increased production of intestinal triglyceride rich lipoproteins in patients with isolated fasting hypertriglyceridemia.

The objective of this study is to compare the serum apoB48 rate after a standardized load test, among patients with isolated hypertriglyceridemia and patients with metabolic syndrome.

DETAILED DESCRIPTION:
Two major studies in 2007 showed that the occurrence of myocardial infarction and death was more frequent in subjects with the highest "non-fasting" triglycerides level. This is an important point that supports the hypothesis that the development of atheromatous lesions also depends on "remnant" of triglyceride-rich lipoproteins (TRL) products such as chylomicrons in the intestine. The elevation of triglycerides in postprandial period depends on the intestinal production of TRL that can be excessively increased as has been shown in diabetes. Accordingly, it is necessary to distinguish between hepatic and intestinal production of TRL in hypertriglyceridemic patients particularly during postprandial period. TRL contain a single molecule of apolipoprotein B (apoB), apoB100 when produced by the liver or apoB-48 when they are produced by the gut. It is well known that apo B100 is the lipoprotein of the VLDL which is increased in hypertriglyceridemia. But preliminary works showed that fasting concentrations of apoB48 were correlated with triglycerides in some hypertriglyceridemic patients. These results suggest an intestinal part in fasting triglycerides levels. It therefore appears that the liver and intestine contribute to hypertriglyceridemia, but the intestinal part is not established particularly in isolated hypertriglyceridemia. The detection of abnormalities in the production of LRT would consider intestinal bowel as a target organ for the initiation of specific lipid-lowering therapy.

ELIGIBILITY:
Inclusion criteria :

1. Patient who provided his consent in writing before the completion of any procedure related to the Protocol
2. Patient affiliated to the French social security system or to another similar insurance
3. Men and women aged from 18 years to 75 years
4. Patient of Department of Endocrinology-Metabolism and hospitalized for a medical checkup
5. Fasting hypertriglyceridemia >1.5 g / L
6. No lipid-lowering treatment or omega 3
7. Patients with an untreated systolic blood pressure <130mmHg and diastolic <85mmHg
8. Stable weight (variation less than 5 kg in the month before inclusion)

Inclusion in the metabolic syndrome group if :

* Fasting glucose > 5.6 mmol / L but <7.0 mmol / L and
* Waist perimeter >94 cm in men and >80cm in women.

Inclusion in isolated hypertriglyceridemia group: patients not having the criteria of the group "metabolic syndrome"

Exclusion criteria :

1. Diabetic Patient
2. Any recent changes (less than one month) of any treatment
3. Patient participating in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Apo B48 plasma concentration | every hour for 6 hours (day of sampling after postprandial test)
  Area under the Apo B48 (g/L) plasma concentration (g/L) measured every hour for 6 hours versus time curve (AUC).

SECONDARY OUTCOMES:
Apo B48 peak plasma concentration | the highest level of Apo B48 during the test of 6 hours (day of sampling after postprandial test)
  Apo B48 (g/L) peak plasma concentration (Cmax)

OTHER OUTCOMES:
Apo B100 plasma concentration | every hour for 6 hours (day of sampling after postprandial test)
  Area under the Apo B100 (g/L) plasma concentration (g/L) measured every hour for 6 hours versus time curve (AUC).
Apo B100 peak plasma concentration | the highest level of Apo B100 during the test of 6 hours
  Apo B100 (g/L) peak plasma concentration (Cmax)
Triglycerides peak plasma concentration | The highest level of triglycerides during the test of 6 hours
  Triglycerides (g/L) peak plasma concentration (Cmax)
Glycemia plasma concentration | every hour for 6 hours
  Area under the glycemia plasma concentration (mmol/L) measured every hour for 6 hours versus time curve (AUC)
Glycemia peak plasma concentration | the highest level of glycemia during the 6-hours postprandial test
  Glycemia (mmol/L/L) peak plasma concentration (Cmax) during the postprandial test

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Giral, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié Salpetriere Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giral P, Simon D, Chapman MJ. Letter by Giral et al regarding article, "lipoprotein(a) concentrations, rosuvastatin therapy, and residual vascular risk: an analysis from the JUPITER trial (justification for the use of statins in prevention: an intervention trial evaluating rosuvastatin)". Circulation. 2014 Oct 21;130(17):e151. doi: 10.1161/CIRCULATIONAHA.114.009590. No abstract available. PMID 25332284